CLINICAL TRIAL: NCT03675568
Title: Non-cultured Autologous Keratinocyte Suspension for Treatment of Deep Dermal Burn and Post-Burn Raw Area Versus Traditional Split Skin Graft
Brief Title: Non-cultured Autologous Keratinocyte Suspension Versus Traditional Split Skin Graft for Burn Wounds Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject changed
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Diefy Salem, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCAKS
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Burn Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Non-Cultured autologous keratinocyte suspension
  Interventions: Procedure: Non-cultured keratinocyte suspension
- Control group (Active Comparator): Split skin Graft
  Interventions: Procedure: Split skin Graft

INTERVENTIONS:
Procedure: Non-cultured keratinocyte suspension — A new method for treatment of burn wounds
  Arms: study group
Procedure: Split skin Graft — A traditional method for treatment of burn wounds
  Arms: Control group

SUMMARY:
A study comparing effect of non-cultured autologous keratinocyte suspension on burn wounds treatment compared with traditional split skin graft

DETAILED DESCRIPTION:
Burn injuries are complicated wounds to manage with a relative high mortality rate in especially large area burns and elderly patients.

Substantial tissue damage and extensive fluid loss can cause impaired vital functions of the skin. When healing is delayed, the potential short term common complications include wound infection affecting the local healing process or systemic inflammatory and immunological responses which subsequently can cause life threatening sepsis and multi-organ failure.

Fortunately, survival rates have improved drastically over the last century due to advancements in burn care such as early surgical intervention, critical care support and wound care.

For many years the "gold standard" for treating wounds of burn patients has been transplantation with an autologous split skin graft. In patients with extensive burn wounds donor sites may be limited. In order to cover all the wounds, the patients often need multiple operations and/or the skin had to be expanded as much as possible.

However, the current different expansion techniques and treatments [mesh and Meek-Wall] frequently lead to scar formation, especially in the large mesh inter-sites.

The rate of wound closure depends on how quickly epidermal cells migrate out of the meshed auto graft and/ or wound edges to close the wound. Accelerating re-epithelialization could potentially improve the outcome of the healing process in terms of reducing granulation tissue formation, reducing the healing time, and thereby reducing the risk of colonization and infection, as well as scar formation.

Since clinical cases were first successfully treated with cultured epithelial layers, keratinocyte sheets have become an important tool in burn wound treatment. However, the clinical application can be limited by long culture time and fragility of the keratinocyte sheets. There is, therefore, a clinical demand for other options to cover large areas of burn wounds in the absence of viable donor sites.

A novel concept consists of treating wounds with epithelial cell suspensions. In 1998, Fraulin et al. developed a method of spreading cell suspension on to wounds using an aerosol spray in a porcine model.

The use of non-cultured keratinocyte suspensions was first reported by Hunyadi et al., showing that a group of patients with burn wounds or chronic leg ulcers, treated with a fibrin matrix containing keratinocytes, healed completely, as opposed to the control group.

In porcine wound models, non-cultured keratinocyte suspensions have been shown to accelerate wound healing, improve quality of epithelialization, and restore melanocyte population, compared to the respective control group.

Major advantages in the use of non-cultured cell suspensions are a drastic reduction of preparation time and possibly easier handling compared to keratinocyte sheets. Particularly, scar quality may be improved by enhancing the speed of epithelialization and fading of mesh patterns in split skin grafts.

In this study, we will compare the results of treating both deep dermal burn wound -following early excision- and post-burn raw area using non-cultured autologous keratinocyte suspension and traditional split skin graft.

ELIGIBILITY:
Inclusion Criteria:

* Deep dermal burns more than 10% total body surface area which require surgical debridement and epidermal replacement.
* Post-burn raw area more than 10% total body surface area

Exclusion Criteria:

* Presence of pre-existing local and systemic bacterial infections.
* Pre-existing medical conditions that would interfere with wound healing (uncontrolled diabetes mellitus, malignancy, congestive heart failure, autoimmune disease, renal failure, corticosteroids and immunosuppressive drugs).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
mean Hospital stay | 1 month
  Number of days patient stays admitted

SECONDARY OUTCOMES:
mean healing time | 1 month
  Number of days until 95% healing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson PC, Hardwicke J, Bamford A, Nightingale P, Wilson Y, Papini R, Moiemen N. Revised estimates of mortality from the Birmingham Burn Centre, 2001-2010: a continuing analysis over 65 years. Ann Surg. 2014 May;259(5):979-84. doi: 10.1097/SLA.0b013e31829160ca. PMID 23598383
- [Background] Osler T, Glance LG, Hosmer DW. Simplified estimates of the probability of death after burn injuries: extending and updating the baux score. J Trauma. 2010 Mar;68(3):690-7. doi: 10.1097/TA.0b013e3181c453b3. PMID 20038856
- [Background] McGwin G Jr, Cross JM, Ford JW, Rue LW 3rd. Long-term trends in mortality according to age among adult burn patients. J Burn Care Rehabil. 2003 Jan-Feb;24(1):21-5. doi: 10.1097/00004630-200301000-00006. PMID 12543987
- [Background] Deitch EA, Wheelahan TM, Rose MP, Clothier J, Cotter J. Hypertrophic burn scars: analysis of variables. J Trauma. 1983 Oct;23(10):895-8. PMID 6632013
- [Background] Hefton JM, Madden MR, Finkelstein JL, Shires GT. Grafting of burn patients with allografts of cultured epidermal cells. Lancet. 1983 Aug 20;2(8347):428-30. doi: 10.1016/s0140-6736(83)90392-6. PMID 6135914
- [Background] Fraulin FO, Bahoric A, Harrop AR, Hiruki T, Clarke HM. Autotransplantation of epithelial cells in the pig via an aerosol vehicle. J Burn Care Rehabil. 1998 Jul-Aug;19(4):337-45. doi: 10.1097/00004630-199807000-00012. PMID 9710733
- [Background] Hunyadi J, Farkas B, Bertenyi C, Olah J, Dobozy A. Keratinocyte grafting: a new means of transplantation for full-thickness wounds. J Dermatol Surg Oncol. 1988 Jan;14(1):75-8. doi: 10.1111/j.1524-4725.1988.tb03343.x. PMID 2447135